CLINICAL TRIAL: NCT00136682
Title: Postoperative Recovery in Patients Receiving Patient-Controlled Epidural Analgesia (PCEA) Compared to Patient-Controlled Intravenous Analgesia (PCA) After Major Open Gynecologic Surgery: A Randomized Controlled Trial
Brief Title: Patient-Controlled Epidural Analgesia (PCEA) for Patients Who Have Had Major Open Gynecologic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Nadeem Abu-Rustum, MD, Memorial Sloan-Kettering Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-091
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-11

CONDITIONS: Postoperative Pain
Keywords: Major abdominal or pelvic surgery; Patient-Controlled Epidural Analgesia (PCEA); Length of hospital stay after surgery
MeSH Terms: conditions — Pain, Postoperative

ARMS (2):
- (PCEA) (Active Comparator): patient-controlled epidural analgesia PCEA involves having an epidural catheter placed before surgery.The epidural catheter will be used during surgery to give drugs, such as morphine and a local anesthetic bupivacaine, which will help control pain. After surgery, a constant flow of pain-reducing medicine, such as morphine, will be given through the catheter. This is controlled by the patient.
  Interventions: Drug: patient-controlled epidural analgesia (PCEA)
- PCA (Active Comparator): patient-controlled intravenous analgesia (PCA) PCA involves placing a tube into the patient's vein after surgery. The tube is connected to a pump that is controlled by the patient. The pump holds a medicine, such as morphine, that eases pain.
  Interventions: Drug: patient-controlled intravenous analgesia (PCA)

INTERVENTIONS:
Drug: patient-controlled epidural analgesia (PCEA) — During the consent process you will be given a patient data sheet to assess your baseline pain and itchiness. While in the hospital you will be given a patient data sheet to fill out information regarding pain, nausea, when you passed gas, and when you ate food. This will be done once a day by a research assistant or by the research investigators.
  Arms: (PCEA)
Drug: patient-controlled intravenous analgesia (PCA) — During the consent process you will be given a patient data sheet to assess your baseline pain and itchiness. While in the hospital you will be given a patient data sheet to fill out information regarding pain, nausea, when you passed gas, and when you ate food. This will be done once a day by a research assistant or by the research investigators.
  Arms: PCA

SUMMARY:
Recovery after major abdominal surgery can be longer than other types of surgery. This is because often after abdominal surgery, the bowel does not work normally. When this happens, patients are unable to pass gas. This can lead to bloating, pain, nausea and vomiting. These symptoms are called postoperative ileus.

We, the researchers at Memorial Sloan-Kettering Cancer Center (MSKCC), are doing this study to compare two methods of treating pain during and after major gynecological surgery. The two methods are called patient-controlled epidural analgesia (PCEA) and patient-controlled intravenous analgesia (PCA). PCA is the standard of care for women having major gynecological surgery. We are going to compare PCEA to PCA to see if PCEA will improve recovery after major gynecologic surgery.

PCEA is a well established method used to ease pain in many settings such as during childbirth and bowel surgery. There have been several studies showing that PCEA is as good as and sometimes better for pain relief than PCA. PCEA may help the bowel work better by preventing ileus after surgery. However, this has never been looked at in women having major gynecologic surgery. This study will also look at whether preventing this ileus will lead to patients going home or returning to regular activities sooner.

DETAILED DESCRIPTION:
The objective of this study is pain at rest and coughing in addition to determine the effect of intraoperative and postoperative thoracic patient-controlled epidural analgesia (PCEA) compared to postoperative intravenous patient-controlled analgesia (PCA) on postoperative recovery parameters, such as time to potential discharge and resumption of intestinal function after major open gynecologic surgery. The population included in this study will be women undergoing a laparotomy for major abdominal or pelvic surgery by the gynecology service. There will be a total of 240 women recruited for this study, with an accrual rate of 5 to 10 patients per month. This study will be a randomized controlled clinical trial. Subjects will be randomized to either general anesthesia with postoperative intravenous patient controlled analgesia (control group) or general anesthesia with intraoperative thoracic epidural anesthesia and postoperative thoracic patient-controlled epidural analgesia (treatment group). This study will not be blinded because of the ethical issues with placing a "sham" epidural catheter in half of the study participants. These patients will be followed prospectively and relevant postoperative parameters will be measured in both groups and compared. This study will address the potential benefits of epidural analgesia on multiple measurements of postoperative recovery. This study will address the potential benefits of epidural analgesia on multiple measurements of postoperative recovery. The primary outcome of interest in this study is pain at rest and when coughing. The secondary outcome is the time to potential discharge.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing a laparotomy for major abdominal or pelvic surgery by the gynecology service
* Patients 18 years or older
* Patients who have signed an approved informed consent form

Exclusion Criteria:

* Patients undergoing total pelvic exenteration
* Patients undergoing laparoscopy only
* Patients undergoing palliative surgery for bowel obstruction
* Patients undergoing emergent operations
* Inability to take oral intake
* Current history of chronic (three months) opioid use or known active alcohol abuse
* Patients with significant cognitive impairment or documented psychologic impairment
* Patients with a history of documented anaphylaxis or contraindication to any of the study medications or standardized intraoperative medications will be excluded from study. These include:

  * Morphine
  * Bupivicaine
* Contraindication to epidural catheter placement. This includes:

  * Documented preoperative coagulopathy: international normalized ratio (INR) < 1.3 and partial thromboplastin time (PTT) < 42
  * Evidence of infection at potential epidural site
  * Prior extensive spinal surgery or major spinal deformity
  * Platelets > 100K (bleeding diatheses, preoperative use of anti-coagulant with planned use of therapeutic dose of anti-coagulant post-operatively)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2004-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pain at rest and when coughing - assessed by visual analog scale (VAS) | conclusion of the study

SECONDARY OUTCOMES:
The time (in days) to potential discharge based on documentation of all of the discharge criteria below: Toleration of diet (as assessed by tolerating clear fluid diet for 24 hours without nausea requiring antiemetic or vomiting within 4 hours of a meal) | conclusion of the study
Passing of flatus (as assessed by patient) | conclusion of the study
Absence of fever for 24 hours | conclusion of the study
Actual length of stay in hospital (in days). This may be different from actual time of potential discharge as met by criteria in primary outcome | conclusion of the study
Nausea (yes/no) | conclusion of the study
Vomiting (number episodes per day) | conclusion of the study
Use of anti-emetics per day (yes/no) | conclusion of the study
Pruritus per day (yes/no) | conclusion of the study
Overall patient satisfaction - questionnaire | conclusion of the study
Postoperative complications - complications occurring within 30 days of surgery as assessed by MSKCC surgical secondary events grading system | conclusion of the study
Complications related to intraoperative events (anesthetic and surgical) | conclusion of the study
Complications arising from analgesic techniques | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem R. Abu-Rustum, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: (Memorial Sloan-Kettering Cancer Center) — http://mskcc.org